CLINICAL TRIAL: NCT01046500
Title: Myo-inositol Versus Metformin Administration in Post-menopausal Women With Metabolic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, Associate Professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INOMEN-2010
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome
Keywords: insulin resistance; body mass index; myo-inositol; serum triglycerides and cholesterol; blood pressure; metformin
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Inositol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator)
  Interventions: Drug: Metformin
- myo-inositol (Active Comparator)
  Interventions: Dietary Supplement: myo-inositol

INTERVENTIONS:
Dietary Supplement: myo-inositol — 2 grams twice a day
  Arms: myo-inositol
Drug: Metformin — pill, 250 mg, twice a day
  Arms: metformin

SUMMARY:
Myo-Inositol is classified as a member of the vitamin B complex. It is a constituent of living cells and is widespread in many food. It is involved in a number of biological processes, including insulin signal transduction, resulting in modulating insulin sensitivity. One hundred post-menopausal women from 50 to 60 years old, affected by metabolic syndrome (criteria are described in NIH ATP III) will be randomized into two groups: 50 treated with myo-inositol 2 g twice per day and fifty treated with metformin for six months. Metformin is the drug usually used in diabetic and pre-diabetic conditions, as metabolic syndrome. The investigators hypothesize that the administration of myo-inositol would improve the insulin-receptor activity in these women, reducing insulin resistance as well as metformin.

OUTCOME MEASURE: HOMA-IR, blood pressure level, serum triglycerides and cholesterol, BMI and waist circumference

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal outpatients affected by the metabolic syndrome, whose criteria are described in NIH ATP III, 2001.

Exclusion Criteria:

* Post-menopausal outpatients without metabolic syndrome
* assumption of hypocholesterolemic or other insulin sensitizing drugs

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
glycaemia, insulinaemia, HOMA-IR | at baseline and after 6 months

SECONDARY OUTCOMES:
serum triglycerides, HDL and total cholesterol, blood pressure level, BMI and waist circumference | at baseline and after six months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Messina, Italy